CLINICAL TRIAL: NCT00077324
Title: Use Of Proteomic Analysis Of Serum Samples For Detection Of Non-Small Cell Lung Cancer
Brief Title: Proteomic Profiling in Diagnosing Non-Small Cell Lung Cancer in Patients Who Are Undergoing Lung Resection for Suspicious Stage I Lung Lesions
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACOSOG-Z4031; CDR0000350123 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Spectrometry, Mass, Matrix-Assisted Laser Desorption-Ionization; Biopsy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgery + blood and serum collection: Patients undergo lung resection. Patients also undergo preoperative and postoperative collection of whole blood and serum for proteomic profiling using surface-enhanced laser desorption/ionization-time of flight mass spectrometry. A lung tissue biopsy taken at surgery is also analyzed.
  Patients are followed at 60-90 days and then annually for 2-5 years.
  Interventions: Genetic: proteomic profiling; Other: surface-enhanced laser desorption/ionization-time of flight mass spectrometry; Procedure: biopsy; Procedure: surgery

INTERVENTIONS:
Genetic: proteomic profiling
Other: surface-enhanced laser desorption/ionization-time of flight mass spectrometry
Procedure: biopsy
Procedure: surgery

SUMMARY:
RATIONALE: Evaluating specific proteins in the blood may be an effective and noninvasive procedure to help doctors determine if a patient has early non-small cell lung cancer.

PURPOSE: This clinical trial is studying proteomic profiling to see how well it works in diagnosing non-small cell lung cancer in patients who are undergoing resection for suspicious (abnormal) stage I lung lesions.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine, prospectively, whether serum proteomic profiling can predict the presence of primary non-small cell lung cancer in patients with clinically suspicious stage I lung lesions who are undergoing lung resection.

Secondary

* Correlate the serum proteomic profile with pathologic nodal status and histopathologic features of primary lung cancer in these patients.
* Correlate the initial and follow-up serum proteomic profile with overall and cancer-specific survival of these patients.
* Correlate changes in the proteomic profile (preoperative to postoperative) with overall and cancer-specific survival of these patients.

Tertiary

* Determine whether novel molecular strategies can predict the presence of lung cancer and/or the biologic behavior of an individual cancer in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be ≥18 years of age.
2. Patient must have a clinically suspicious stage I (cT1-2 N0 M0) lung lesion.
3. Patient must have pre-operative imaging procedures within 60 days prior to the date of the lung resection: Helical CT scan of the chest and CT scan of the upper abdomen, including the liver and adrenal glands (with or without IV contrast), as clinically indicated. The helical CT must rule out metastatic disease in the liver and adrenal glands.
4. Patient, or the patient's legally acceptable representative, must provide a signed and dated written informed consent PRIOR to registration and any study-related procedures being performed.
5. Patient must provide written authorization to allow the use and disclosure of their protected health information. NOTE: This may be obtained in either the study-specific informed consent or in a separate authorization form and must be obtained from the patient PRIOR to registration and any study-related procedures being performed.
6. If patient is a survivor of a prior cancer, the following criteria are met:

   1. Patient has undergone potentially curative therapy for all prior malignancies,
   2. No evidence of any prior malignancies for at least 5 years with no evidence of recurrence (except for effectively treated basal cell or squamous carcinoma of the skin, carcinoma in-situ of the cervix that has been effectively treated by surgery alone, or lobular carcinoma in-situ of the ipsilateral or contralateral breast treated by surgery alone),
   3. Patient is deemed by their treating physician to be at low risk for recurrence from prior malignancies.

Exclusion Criteria:

1. Patient has undergone previous lung resection within the preceding 30 days.
2. Patient has received prior chemotherapy or radiotherapy.
3. Patient has had a blood product transfusion of any kind within the past 60 days of the operative procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2004-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Determine whether the serum proteomic profile can predict the presence of primary lung cancer in patients with suspicious lung lesions | Up to 5 years
Survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David H. Harpole, MD, Study Chair — Duke Cancer Institute
Locations (73):
- United States (72):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - John Muir/Mount Diablo Cancer Center - Concord Campus, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Veterans Affairs Medical Center - Loma Linda (Pettis), Loma Linda, California
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - Praxair Cancer Center at Danbury Hospital, Danbury, Connecticut
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Winship Cancer Institute of Emory University, Altanta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - Jewish Hospital, Louisville, Kentucky
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Fox Chase Cancer Center at St. Francis Medical Center, Trenton, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Benedictine Hospital, Kingston, New York
  - South Nassau Communities Hospital, Oceanside, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Cancer Treatment Center at Good Samaritan Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Jameson Memorial Hospital - North Campus, New Castle, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - U.T. Cancer Institute at University of Tennessee Medical Center, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - LDS Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Harpole DH, Meyerson SL. Lung cancer staging: proteomics. Thorac Surg Clin. 2006 Nov;16(4):339-43. doi: 10.1016/j.thorsurg.2006.10.001. PMID 17240821
- [Result] Grogan EL, Deppen SA, Ballman KV, et al.: Accuracy of FDG-PET to diagnose lung cancer in the ACOSOG Z4031 trial. [Abstract] J Clin Oncol 30 (Suppl 15): A-7008, 2012.
- [Result] Harpole D, Ballman KV, Oberg AL, et al.: Proteomic analysis for detection of NSCLC: results of ACOSOG Z4031. [Abstract] J Clin Oncol 29 (Suppl 15): A-7003, 2011.